CLINICAL TRIAL: NCT01487720
Title: A Prosepctive Phase II Study of Gemcitabine and Oxaliplatin in Combination With Prednisolone for the Treatment of Hormone Refracotry Metastatic Prostate Cancer Previously Treated With Docetaxel Regimen
Brief Title: GEMOX in Docetaxel-Refractory Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, JLee, Associate Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UOSG-AMC-0802
Record Dates: First submitted 2011-12-06; First posted 2011-12-07 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-11

CONDITIONS: Prostate Cancer
Keywords: Castration-resistant prostate cancer; Docetaxel-refractory status
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GEMOX (Experimental): GEMOX treatment
  Interventions: Drug: GEMOX

INTERVENTIONS:
Drug: GEMOX — Gemcitabine 1000 mg/m2 IV on day 1 every 2 weeks (fixed-dose rate 10 mg/m2/min) Oxaliplatin 100 mg/m2 IV on day 1 every 2 weeks Prednisolone 5 mg twice a day orally daily

SUMMARY:
Prostate cancer is one of the most common malignancies affecting men all over the World. Metastatic prostate cancer responds to androgen deprivation for a variable period (20-25 months). Prostate cancer that grows despite castrate levels of testosterone and that no longer responds to any form of hormonal manipulation is defined as castrate resistant prostate cancer (CRPC).

Docetaxel combined with prednisolone has been shown to not only improve QOL and PSA response in CRPC, but also extend the overall survival1. However, the efficacy of the drug has not been universally effective, and nearly all patients have disease progression after docetaxel treatment.

After failure of a docetaxel regimen, With the exception of cabazitaxel or abiraterone, which are not widely and easily availabe in Korea, little treatment regimen can be applied to the patients with reasonable response and benefits.

Gemcitabine is a nucleoside analog with activity against a broad spectrum of solid tumors. When gemcitabine is used as first-line therapy for CRPC, disease control rate was 33% with median duration of 7.1 months. When it is combined with prednisone and zoledronic acid in pretreated patients with CRPC, the PSA response rate was 23% with a disease control rate of 57% in patients with measurable disease.

Oxaliplatin is newer platinum agent that has favorable toxicity profile and evidence of activity in cisplatin-resistant cell lines. Droz et al. performed a multicenter phase II study in 54 patients with metastatic CRPC who were randomized to receive oxaliplatin either alone or with 5-FU. More than 50% of the patients had received prior chemotherapy including cisplatin. Despite heavy pretreatment, PSA desclines were noted in 11% and 19% of patients in each arm.

Gemcitabine plus oxaliplatin combination was widely studied and has been reported to be safe and effective in various cancers.

This study is to assess the efficacy and safety of GEMOX in docetaxel-refractory CRPC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Clinical or radiologic evidence of metastatic disease
* Documented disease progression during hormone therapy (ADT plus antiandrogen) and no response to ADT withdrawal
* Docetaxel-refractory disease defined as disease progression documented either during treatment of within 60 days after the cessation of treatment with docetaxel
* Prior exposure to estramustine or mitoxantrone is allowed
* KPS ≥ 60
* No prior radioisotope therapy
* No prior radiotherapy 25% or more of the bone marrow
* No peripheral neuropathy grade 2 or worse
* Adequate organ and bone marrow function

Exclusion Criteria:

* Other tumor type than adenocarcinoma
* Presence or history of CNS metastasis
* Other serious illness or medical conditions

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
PSA response | 6 months
  Based on PCWG 1.0

SECONDARY OUTCOMES:
PSA decline | 6 months
  Based on PCWG 2.0
Time to PSA progression | 12 months
Composite progression-free survival | 12 months
  Based on RECIST, bone scan, and performance status
RECIST Response | 6 months
  Based on RECIST v 1.1
Safety | 6 months
  Based on NCI CTCAE v. 4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea